CLINICAL TRIAL: NCT00433381
Title: A Randomized Phase II Trial of Bevacizumab With Irinotecan or Bevacizumab With Temozolomide in Recurrent Glioblastoma
Brief Title: Bevacizumab and Irinotecan or Temozolomide in Treating Patients With Recurrent or Refractory Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: American College of Radiology Imaging Network (Network); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00743; NCI-2009-00743 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-0625 (Other: RTOG); ACRIN-6677 (Other: ACRIN); CDR0000528259 (Registry Identifier: CDR); RTOG 0625 (Other: Radiation Therapy Oncology Group); RTOG-0625 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-08

CONDITIONS: Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Irinotecan; Temozolomide

ARMS (2):
- Arm I (bevacizumab and temozolomide) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral temozolomide once daily on days 1-21.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide
- Arm II (bevacizumab & irinotecan hydrochloride) (Experimental): Patients receive bevacizumab IV as in Arm I followed by irinotecan hydrochloride IV over 90 minutes on days 1 and 15.
  Interventions: Biological: Bevacizumab; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
  Arms: Arm II (bevacizumab & irinotecan hydrochloride)
Drug: Temozolomide — Given orally
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac
  Arms: Arm I (bevacizumab and temozolomide)

SUMMARY:
This randomized phase II trial is studying the side effects and how well giving bevacizumab together with irinotecan or temozolomide works in treating patients with recurrent or refractory glioblastoma multiforme or gliosarcoma. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with irinotecan or temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of bevacizumab and irinotecan hydrochloride, in terms of 6-month progression-free survival rate, in patients with recurrent or refractory intracranial glioblastoma multiforme or gliosarcoma.

II. Determine the adverse event profile and tolerability of bevacizumab and temozolomide in these patients.

SECONDARY OBJECTIVES:

I. Determine the efficacy of bevacizumab and temozolomide, in terms of 6-month progression-free survival rate, in patients previously treated with temozolomide.

II. Determine the efficacy of bevacizumab and irinotecan hydrochloride, in terms of objective response, in patients with measurable disease.

III. Determine the efficacy of bevacizumab and temozolomide, in terms of objective response, in patients with measurable disease who were previously treated with temozolomide.

IV. Determine the toxicity profile and tolerability of bevacizumab and irinotecan hydrochloride in these patients.

TERTIARY OBJECTIVES:

I. Assess the potential role of perfusion MRI and magnetic resonance spectroscopy imaging as an early indicator of response to therapy after 2 weeks of treatment with bevacizumab.

II. Assess the potential role of perfusion MRI and magnetic resonance spectroscopy imaging as a prognostic indicator based on images taken at baseline, at 2 weeks, and after 2 courses of study treatment.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (< 50 vs >= 50 years of age) and Karnofsky performance status (70-80% vs 90-100%). Patients are randomized to 1 of 2 treatment arms with a 2:1 ratio (arm I:arm II).

ARM I: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral temozolomide once daily on days 1-21.

ARM II: Patients receive bevacizumab IV as in Arm I followed by irinotecan hydrochloride IV over 90 minutes on days 1 and 15.

In both arms, treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. All patients undergo MRI at baseline and at every 2 courses (no 2-week MRI) per standard of care until progression or discontinuation of treatment to assess areas of breakdown of the blood-brain barrier. Patients undergo an additional MRI after study therapy. Consenting patients also undergo diffusion and perfusion MRI and magnetic resonance spectroscopic imaging for correlative studies.

After completion of study therapy, patients are followed up for at least 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intracranial glioblastoma multiforme (GBM) or gliosarcoma

  * Original histology of low-grade glioma with subsequent histological diagnosis of GBM or gliosarcoma allowed
* Recurrent or refractory disease, meeting all of the following criteria:

  * Must have received prior temozolomide
  * Pathologic or imaging confirmation of tumor progression or regrowth required

    * Confirmation of true progressive disease (rather than radiation necrosis) by positron emission tomography, thallium scanning, MRI spectroscopy, or surgical documentation required for patients who received prior interstitial brachytherapy, Gliadel wafer, or stereotactic radiosurgery
* Unequivocal radiographic evidence of tumor progression by MRI within the past 14 days (while on a stable dose of steroids for ? 5 days)
* No acute intratumoral hemorrhage on MRI

  * Patients with MRI demonstrating old hemorrhage or subacute blood after a neurosurgical procedure (biopsy or resection) are eligible
* Karnofsky performance status 70-100%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after completion of bevacizumab therapy
* Systolic blood pressure ? 160 mm Hg or diastolic blood pressure ? 90 mm Hg (antihypertensive medication allowed)
* Able to undergo brain MRI scans with intravenous gadolinium
* Absolute neutrophil count ? 1,500 cells/mm?
* Platelet count ? 100,000 cells/mm?
* Hemoglobin ? 10 g/dL (transfusion or other intervention allowed)
* WBC ? 3,000 cells/mm?
* AST < 2 times upper limit of normal
* Bilirubin ? 1.6 mg/dL
* Creatinine < 1.5 mg/dL
* Urine protein:creatinine ratio ? 0.5 by urinalysis OR total urinary protein < 1,000 mg by 24-hour urine collection
* INR < 1.4 (for patients not on warfarin)
* No patients with severely impaired renal function (i.e., estimated glomerular filtration rate < 30 mL/min or on dialysis)
* No other prior invasive malignancy, except nonmelanomatous skin cancer or carcinoma in situ of the cervix, unless the patient has been disease free and off therapy for that disease for ? 3 years
* No severe, active comorbidity, defined as any of the following:

  * Transmural myocardial infarction or unstable angina within the past 6 months
  * Evidence of recent myocardial infarction or ischemia manifested as ST elevation of ? 2 mm by EKG performed within the past 14 days
  * New York Heart Association class II-IV congestive heart failure requiring hospitalization within the past 12 months
  * History of stroke or transient ischemic attack within the past 6 months
  * Cerebrovascular accident within the past 6 months
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g., aortic aneurysm or history of aortic dissection)
  * Clinically significant peripheral vascular disease
  * Evidence of bleeding diathesis or coagulopathy
  * Serious or nonhealing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study entry
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within the past 14 days
  * Acquired immune deficiency syndrome (AIDS)
* No significant traumatic injury within the past 28 days
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No condition that impairs the ability to swallow pills (e.g., gastrointestinal tract disease resulting in an inability to take oral medication; requirement for IV alimentation; prior surgical procedures affecting absorption; or active peptic ulcer disease)
* No disease that would obscure toxicity or dangerously alter drug metabolism
* No concurrent major surgical procedures
* Recovered from prior therapy
* Recent resection of recurrent or progressive tumor allowed provided the following criteria are met:

  * Failed prior radiotherapy that was completed ? 42 days ago
  * Residual disease after resection of recurrent glioblastoma is not mandated
* More than 28 days since prior surgery or open biopsy
* More than 7 days since prior core or needle biopsy
* At least 28 days since prior investigational agents
* At least 14 days since prior vincristine
* At least 42 days since prior nitrosoureas
* At least 21 days since prior procarbazine
* At least 28 days since other prior cytotoxic therapy
* At least 7 days since prior noncytotoxic agents (e.g., interferon, tamoxifen, thalidomide, or isotretinoin [except radiosensitizers])
* At least 14 days since prior enzyme-inducing antiepileptic drugs (EIAEDs)

  * Concurrent non-hepatic EIAEDs allowed
* No other concurrent CYP3A4 inducers, such as rifampin or Hypericum perforatum (St. John's wort)
* Concurrent full-dose anticoagulants (e.g., warfarin or low molecular weight heparin) allowed provided all of the following criteria are met:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  * In-range INR (usually between 2 and 3) on a stable dose of oral anticoagulants or on a stable dose of low molecular weight heparin
* No concurrent highly active antiretroviral therapy
* No concurrent prophylactic use of growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2010-01-21 (Actual); Study Completion 2011-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gilbert, Principal Investigator — Radiation Therapy Oncology Group
Locations (93):
- United States (93):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Marin General Hospital, Greenbrae, California
  - Sutter Cancer Research Consortium, Novato, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Yale University, New Haven, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - John F Kennedy Medical Center, Edison, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Radiation Therapy Oncology Group, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Saint Francis Hospital, Federal Way, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Bevacizumab and Temozolomide): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral temozolomide once daily on days 1-21 of a 28-day cycle. Up to 24 cycles for patients demonstrating evidence of benefit as defined by stable or responding tumor.
- Arm II (Bevacizumab and Irinotecan Hydrochloride): Patients receive bevacizumab IV as in Arm I followed by irinotecan hydrochloride IV over 90 minutes on days 1 and 15 of a 28-day cycle. Up to 24 cycles for patients demonstrating evidence of benefit as defined by stable or responding tumor.
Period: Overall Study
Arm/Group | Arm I (Bevacizumab and Temozolomide) | Arm II (Bevacizumab and Irinotecan Hydrochloride)
Started | 63 | 60
Completed | 60 (Subjects contributing data to [the primary] analysis are considered to have completed the study.) | 57
Not Completed | 3 | 3
Not completed — Ineligible / no protocol treatment | 3 | 3

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Bevacizumab and Temozolomide) | Arm II (Bevacizumab and Irinotecan Hydrochloride) | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Continuous [Median (Full Range); unit: years] | 57.5 [24 to 82] | 55 [23 to 78] | 56 [23 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Count/Percentage of Patients Progression-free at 6 Months for Bevacizumab and Irinotecan Hydrochloride Arm
Description: Progression defined as ≥ 25% increase in the size of enhancing tumor or any new tumor; or neurologically worse, and steroids stable or increased. Percentage is calculated by taking the number of patients who have survived 6 months without progression of study disease after study registration in the numerator. The denominator consists of all patients except those who were found retrospectively to be ineligible or who were lost to follow-up after less than 6 months.
Time Frame: From randomization to six months.
Population: Eligible patients with six-month data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (Bevacizumab and Irinotecan Hydrochloride)
Number analyzed (Participants) | 57
Participants | 22
Statistical Analysis 1: Comparison: Arm II (Bevacizumab and Irinotecan Hydrochloride); Null hypothesis: 20% of patients progression-free at six months. Alternative hypothesis: 35%. Type I and II error rates = 0.10. Required sample size = 57; Test type: Other; The determination of treatment efficacy was to be made made based on the following rules: If 16 or more of the cases (16/57=28.1%) are progression free and alive at 6 months, then reject the null hypothesis that the rate is no better than 20%. If 15 or fewer of the cases (15/57=26.3%) are progression free and alive at 6 months, then reject the alternative hypothesis that the rate is at least 35%

2. Primary Outcome: Count/Percentage of Patients Discontinuing Treatment Due to Treatment-related Medical Complications(Bevacizumab and Temozolomide Arm)
Description: This endpoint determines tolerability of this treatment arm. If tolerable, then the secondary endpoint of treatment efficacy for this arm occurs. Percentage is calculated by taking the number of patients who did not stop bevacizumab and temozolomide treatment due to medical complications in the numerator. The denominator consists of all patients except those who were found retrospectively to be ineligible or who did not begin treatment.
Time Frame: From randomization to end of treatment (treatment can continue up to 24 months for patients with stable or responding tumor).
Population: The first 29 eligible patients who received protocol treatment were to be evaluated for treatment tolerability.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Bevacizumab and Temozolomide)
Number analyzed (Participants) | 29
Participants | 6
Statistical Analysis 1: Comparison: Arm I (Bevacizumab and Temozolomide); Null hypothesis: 35% discontinuation rate of bevacizumab and temozolomide. Alternative hypothesis: 5%. Type I and II error rates = 0.10. Sample size = 29; Test type: Other; The determination of treatment tolerability was to be made based on the following rules: If 6 or fewer of the cases (6/29=20.6%) stop treatment due to medical conditions, then reject the null hypothesis that the discontinuation rate is at least 35% and conclude tolerability. If 7 or more of the cases (7/29=24.1%) stop treatment due to medical conditions, then reject the alternative hypothesis that the discontinuation rate no more than 15%

3. Primary Outcome: Number of Participants With Predicted Progression-free Survival at 6 Months (PFS-6)
Description: Magnetic Resonance Imaging with Spectroscopy (MRS or MRSI) metabolic tumor ratios will be used to predict 6-month progression-free survival (PFS-6) over all study participants. Ratios of NAA/Cho, Cho/Cr, NAA/Cr measured at 2 weeks and 8 weeks and every 2 months until 96wks were used to predict survival, and time to progression, evaluated at 96wks, is the determinate of PFS at 6months (PFS-6). Subjects will not be analyzed by arm.
Time Frame: 2 and 8 weeks posttreatment, and every 2 months until 96wks
Population: A subset of 3 institutions conducted a substudy of advanced MRI, including dynamic contrast enhanced imaging, dynamic susceptibility contrast imaging, and MRSI.
  Of 123 main subjects, a subset of 20 consented to the MRS substudy, of whom 13 had analyzable MRS datasets. this subset is independent of Study Arm.
Measure: Count of Participants; unit: Participants
Groups:
- Analyzable MRS Participants: The subset of 13 participants from any arm with analyzable MRS datasets from the group of 20 who consented to the MRS substudy.
Arm/Group | Analyzable MRS Participants
Number analyzed (Participants) | 13
Participants
  PFS <= 6mo | 4
  PFS > 6mo | 9
Statistical Analysis 1: Comparison: Analyzable MRS Participants; Accuracy estimate, as measured by the Area under the Curve (AUC), for the prediction of PFS-6 by change in metabolic ratio of tumor NAA/Cho at 2 weeks; Test type: Other — Receiver Operating Characteristic (ROC) analysis; Area Under the Curve (AUC) = 0.50, 95% CI 2-sided [0.09 to 0.91]
Statistical Analysis 2: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor Cho/Cr at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.54, 95% CI 2-sided [0.14 to 0.95]
Statistical Analysis 3: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor NAA/Cr at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.46, 95% CI 2-sided [0 to 0.99]
Statistical Analysis 4: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor NAA/Cho at 8 weeks; Test type: Other; Area Under the Curve (AUC) = 0.85, 95% CI 2-sided [0.53 to 1]
Statistical Analysis 5: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor Cho/Cr at 8 weeks; Test type: Other; Area Under the Curve (AUC) = 0.83, 95% CI 2-sided [0.47 to 1]
Statistical Analysis 6: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor NAA/Cr at 8 weeks; Test type: Other; Area Under the Curve (AUC) = 0.60, 95% CI 2-sided [0.11 to 1]
Statistical Analysis 7: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor NAA/Cho at 16 weeks; Test type: Other; Area Under the Curve (AUC) = 0.75, 95% CI 2-sided [0.21 to 1]
Statistical Analysis 8: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor Cho/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 1.0, 95% CI 2-sided [1 to 1]
Statistical Analysis 9: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of tumor NAA/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.46, 95% CI 2-sided [0 to 1]
Statistical Analysis 10: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery NAA/Cho at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.39, 95% CI 2-sided [0 to 0.88]
Statistical Analysis 11: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery Cho/Cr at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.52, 95% CI 2-sided [0.13 to 0.91]
Statistical Analysis 12: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery NAA/Cr at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.54, 95% CI 2-sided [0.06 to 1]
Statistical Analysis 13: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery NAA/Cho at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.47, 95% CI 2-sided [0.02 to 0.92]
Statistical Analysis 14: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery Cho/Cr at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.41, 95% CI 2-sided [0.01 to 0.80]
Statistical Analysis 15: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery NAA/Cr at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.63, 95% CI 2-sided [0.22 to 1]
Statistical Analysis 16: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery NAA/Cho at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 1.00, 95% CI 2-sided [1 to 1]
Statistical Analysis 17: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery Cho/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 1.00, 95% CI 2-sided [1 to 1]
Statistical Analysis 18: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of PFS-6 by change in metabolic ratio of periphery NAA/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.93, 95% CI 2-sided [0.73 to 1]

4. Primary Outcome: Number of Participants With Predicted Overall Survival (OS) at 12 Months
Description: Magnetic Resonance Imaging with Spectroscopy (MRS or MRSI) metabolic tumor ratios will be used to predict 12-month overall survival (OS).
  Ratios of NAA/Cho, Cho/Cr, NAA/Cr measured at 2 weeks and 8 weeks and every 2 months until 96wks were used to predict survival, and time to death, evaluated at 96wks, is the determinate of OS at 12 months. Subjects will not be analyzed by arm.
Time Frame: 2 and 8 weeks posttreatment, and every 2 months until 96wks
Population: A subset of 3 institutions conducted a substudy of advanced MRI, including dynamic contrast enhanced imaging, dynamic susceptibility contrast imaging, and MRSI. Subjects participated in the MR substudies regardless of therapeutic intervention
Measure: Count of Participants; unit: Participants
Groups:
- Analyzable MRS Participants: The subset of 13 participants with analyzable MRS datasets from the 20 who consented to the MRS substudy
Arm/Group | Analyzable MRS Participants
Number analyzed (Participants) | 13
Participants
  OS <=12mo | 6
  OS>12 mo | 7
Statistical Analysis 1: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor NAA/Cho at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.42, 95% CI 2-sided [0 to 0.92]
Statistical Analysis 2: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor Cho/Cr at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.42, 95% CI 2-sided [0 to 0.88]
Statistical Analysis 3: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor NAA/Cr at 2 weeks; Test type: Other — ROC analysis; Accuracy: Area Under the ROC = 0.67, 95% CI 2-sided [0.25 to 1]
Statistical Analysis 4: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor NAA/Cho at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.80, 95% CI 2-sided [0.47 to 1]
Statistical Analysis 5: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor Cho/Cr at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.78, 95% CI 2-sided [0.44 to 1]
Statistical Analysis 6: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor NAA/Cr at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.60, 95% CI 2-sided [0.17 to 1]
Statistical Analysis 7: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor NAA/Cho at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.80, 95% CI 2-sided [0.45 to 1]
Statistical Analysis 8: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor Cho/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.73, 95% CI 2-sided [0.19 to 1]
Statistical Analysis 9: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of tumor NAA/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.57, 95% CI 2-sided [0.03 to 1]
Statistical Analysis 10: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery NAA/Cho at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.60, 95% CI 2-sided [0.20 to 1]
Statistical Analysis 11: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery Cho/Cr at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.72, 95% CI 2-sided [0.36 to 1]
Statistical Analysis 12: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery NAA/Cr at 2 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.50, 95% CI 2-sided [0.06 to 0.94]
Statistical Analysis 13: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery NAA/Cho at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.58, 95% CI 2-sided [0.22 to 0.95]
Statistical Analysis 14: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery Cho/Cr at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.50, 95% CI 2-sided [0.13 to 0.87]
Statistical Analysis 15: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery NAA/Cr at 8 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.78, 95% CI 2-sided [0.47 to 1]
Statistical Analysis 16: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery NAA/Cho at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 1.00, 95% CI 2-sided [1 to 1]
Statistical Analysis 17: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery Cho/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 0.89, 95% CI 2-sided [0.63 to 1]
Statistical Analysis 18: Comparison: Analyzable MRS Participants; AUC (Accuracy) estimate for the prediction of 12 month overall survival by change in metabolic ratio of periphery NAA/Cr at 16 weeks; Test type: Other — ROC analysis; Area Under the Curve (AUC) = 1.00, 95% CI 2-sided [1 to 1]

5. Secondary Outcome: Count/Percentage of Patients Progression-free at 6 Months for Bevacizumab and Temozolomide Arm
Description: as for outcome 1
Time Frame: From randomization to six months.
Population: Eligible patients with six-month data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Bevacizumab and Temozolomide)
Number analyzed (Participants) | 59
Participants | 23
Statistical Analysis 1: Comparison: Arm I (Bevacizumab and Temozolomide); Test type: Other; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Patients' Best Objective Response (Complete Response, Partial Response, Stable Disease, Progression)
Description: Tumor size measured in millimeters and is the largest crosssectional area using perpendicular measurements of contrast enhancing abnormality. Complete response (CR): Complete disappearance of all enhancing tumor on consecutive MRI scans at least 1 month apart, off corticosteroids, and neurologically stable or improved. Partial response (PR): ≥ 50% decrease in size of enhancing tumor on consecutive MRI scans at least 1 month apart, corticosteroids stable or reduced, and neurologically stable or improved. Progressive disease (PD): ≥ 25% increase in the size of enhancing tumor or any new tumor; or neurologically worse, and steroids stable or increased. Stable disease (SD): Does not qualify for CR, PR, or PD.
Time Frame: From randomization to death or last follow-up. Patients were followed up to 62.9 months.
Population: Eligible patients with measurable disease at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Bevacizumab and Temozolomide) | Arm II (Bevacizumab and Irinotecan Hydrochloride)
Number analyzed (Participants) | 58 | 54
Participants
  Complete Response | 2 | 2
  Partial Response | 9 | 13
  Stable Disease | 32 | 26
  Progressive Disease | 10 | 12
  Indeterminate | 5 | 1

7. Secondary Outcome: Agreement Between Local Interpretation and Central Interpretation of Standard MRI
Description: Local and central interpretations of the standard MRI were assessed for progression and survival at all available imaging (baseline visit, week 2, and after every 2 cycles of treatment, and at termination of treatment). Patients who suffer clinical progression without radiographic confirmation of progression were considered to have progressive disease in determination of PFS-6. Subjects participated in the MR substudies regardless of therapeutic intervention
Time Frame: baseline visit, week 2, after every 2 cycles of treatment, and at termination of treatment
Population: Of the 123 subject accrued to ACRIN 6677, 103 were analyzable for this aim. Reasons for exclusions were as follows: 11 subjects only had baseline imaging, 4 were ineligible, 1 was lost to followup, and 4 had incomplete/uninterpretable images.
Measure: Count of Participants; unit: Participants
Groups:
- Standard MRI Local and Central Evaluation: 103 cases with both a central and local interpretation of the standard MRI
Arm/Group | Standard MRI Local and Central Evaluation
Number analyzed (Participants) | 103
Participants
  Local Read: PFS <= 6mo | 62
  Local Read: PFS >= 6mo | 41
  Central Read: PFS <= 6mo | 55
  Central Read: PFS >= 6mo | 48
Statistical Analysis 1: Comparison: Standard MRI Local and Central Evaluation; Agreement between Local and Central determinations 6-month PFS, based on imaging, was evaluated using Kappa statistics; Test type: Other — Agreement was assessed using a Kappa statistic; Kappa Statistic = 0.39, 95% CI 2-sided [0.21 to 0.57]

8. Secondary Outcome: Accuracy of Local PFS 6-mo Interpretation Using Central Review PFS-6 as the Reference Standard
Description: Local reads were treated as the test and central reads were treated as the reference standard. Thus, a participant meeting the definition of progression on any standard MRI central interpretation (baseline visit, week 2, after every 2 cycles of treatment, and at termination of treatment) was considered positive for PFS-6. Therefore, a true positive is defined as a positive local interpretation for a subject with a positive central read.
Time Frame: baseline visit, week 2, after every 2 cycles of treatment, and at termination of treatment
Population: Standard of care MRI occurred at baseline, after every 2 cycles of treatment (every 8 weeks), and after completion/termination of treatment. Subjects participated in the MR substudies regardless of therapeutic intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Standard MRI Local and Central Evaluation
Number analyzed (Participants) | 103
Participants
  Local Read (Test): PFS-6 Negative | 62
  Local Read (Test): PFS-6 Positive | 41
  Central Read (Reference): PFS-6 Negative | 48
  Central Read (Reference): PFS-6 Positive | 55
Statistical Analysis 1: Comparison: Standard MRI Local and Central Evaluation; Sensitivity; Test type: Other — Sensitivity; Sensitivity = 0.6, 95% CI 2-sided [0.46 to 0.73]
Statistical Analysis 2: Comparison: Standard MRI Local and Central Evaluation; Specificity; Test type: Other — Specificity; Specificity = 0.78, 95% CI 2-sided [0.66 to 0.87]

9. Secondary Outcome: Correlation of Degree of Cerebral Blood Volume (CBV) and Lactate (Lac) to N-acetylaspartate (NAA) (Lac/NAA) Ratio
Description: Aim not included in final (February 10, 2009) protocol (removed from section 2).
Time Frame: 2 weeks following initiation of protocol treatment (T1) and at 8 weeks following chemotherapy with bevacizumab (T2)
Population: This Aim was removed from the approved protocol aims. Data were not collected.
Groups:
- No Particpants: This is a NULL group set to represent a population of 0 participants.
Arm/Group | No Particpants
Number analyzed (Participants) | 0

10. Secondary Outcome: Correlation of Degree of Cerebral Blood Volume (CBV) and Lactate (Lac) to Patient Response
Description: Aim not included in final (February 10, 2009) protocol (removed from section 2)
Time Frame: 2 weeks following initiation of protocol treatment (T1)
Population: This Aim was removed from the approved protocol aims. Data were not collected.
Arm/Group | No Particpants
Number analyzed (Participants) | 0

11. Secondary Outcome: Predictive Value of CBV and Lac/NAA in Assessing 6-month Progression-free Survival
Description: Aim not included in final (February 10, 2009) protocol (removed from section 2)
Time Frame: 2 weeks following initiation of protocol treatment (T1)
Population: This Aim was removed from the approved protocol aims. Data were not collected.
Arm/Group | No Particpants
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Perfusion MRI Markers at Week 2 as Predictors of 12mo Overall Survival (OS)
Description: To assess the potential role of perfusion MRI as a prognostic indicator for 12-month OS based on the change in MRI markers evaluated before treatment and 2 weeks following initiation of protocol treatment. Percent change in mean tumor relative cerebral blood volume (rCBV) derived from dynamic susceptibility contrast (DSC) MRI normalized to white matter (nRCBV) and standardized rCBV (sRCBV) between baseline and week 2 are the prognostic indicators.
Time Frame: Baseline and 2 Weeks
Population: Analyzable participants are defined as those participants with DSC data supplied for the baseline scan and at least one scan post-baseline. Subjects participated in the MR substudies regardless of therapeutic intervention
Measure: Number (95% Confidence Interval); unit: Area Under the Curve (AUC)
Groups:
- DSC 2-week Participants: The subset of 13 participants with a baseline and 2-week DSC MRI, from the group of 21 participants with analyzable DSC scans, defined as having both the baseline scan and at least one post-baseline scan that produced usable DSC data
Arm/Group | DSC 2-week Participants
Number analyzed (Participants) | 13
Area Under the Curve (AUC)
  nRCBV (%change @ week2) | 0.85 [0.624 to 1]
  sRCBV (%change @ week2) | 0.825 [0.577 to 1]

13. Secondary Outcome: Change in Perfusion MRI Markers at Week 8 as Predictors of 12mo Overall Survival (OS)
Description: To assess the potential role of perfusion MRI as a prognostic indicator for 12-month OS based on the change in MRI markers evaluated before treatment and 8 weeks following initiation of protocol treatment. Percent change in mean tumor relative cerebral blood volume (rCBV) derived from dynamic susceptibility contrast (DSC) MRI normalized to white matter (nRCBV) and standardized rCBV (sRCBV) between baseline and week 8 are the prognostic indicators.
Time Frame: Baseline and 8 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Area Under the Curve (AUC)
Groups:
- DSC 8-week Participants: The subset of 17 participants with a baseline and 8-week DSC MRI, from the group of 21 participants with analyzable DSC scans, defined as having both the baseline scan and at least one post-baseline scan that produced usable DSC data
Arm/Group | DSC 8-week Participants
Number analyzed (Participants) | 17
Area Under the Curve (AUC)
  nRCBV (%change @ week8) | 0.470 [0.171 to 0.768]
  sRCBV (%change @ week8) | 0.561 [0.277 to 0.844]

14. Secondary Outcome: Change in Perfusion MRI Markers at Week 16 as Predictors of 12mo Overall Survival (OS)
Description: To assess the potential role of perfusion MRI as a prognostic indicator for 12-month OS based on the change in MRI markers evaluated before treatment and 16 weeks following initiation of protocol treatment. Percent change in mean tumor relative cerebral blood volume (rCBV) derived from dynamic susceptibility contrast (DSC) MRI normalized to white matter (nRCBV) and standardized rCBV (sRCBV) between baseline and week 16 are the prognostic indicators.
Time Frame: Baseline and 16 Weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Area Under the Curve (AUC)
Groups:
- DSC 16-week Participants: The subset of 13 participants with a baseline and 16-week DSC MRI, from the group of 21 participants with analyzable DSC scans, defined as having both the baseline scan and at least one post-baseline scan that produced usable DSC data
Arm/Group | DSC 16-week Participants
Number analyzed (Participants) | 13
Area Under the Curve (AUC)
  nRCBV (%change @ week16) | 0.762 [0.435 to 1]
  sRCBV (%change @ week16) | 0.905 [0.736 to 1]

ADVERSE EVENTS:
Description: Eligible patients with adverse event data are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Groups:
- Arm I (Bevacizumab and Temozolomide): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral temozolomide once daily on days 1-21 of a 28-day cycle. Up to 24 cycles for patients demonstrating evidence of benefit as defined by stable or responding tumor. Data is reported for eligible patients with adverse event data who started study treatment, which is 60.
- Arm II (Bevacizumab and Irinotecan Hydrochloride): Patients receive bevacizumab IV as in Arm I followed by irinotecan hydrochloride IV over 90 minutes on days 1 and 15 of a 28-day cycle. Up to 24 cycles for patients demonstrating evidence of benefit as defined by stable or responding tumor. Data is reported for eligible patients with adverse event data who started study treatment, which is 57 patients.
Arm/Group | Arm I (Bevacizumab and Temozolomide) | Arm II (Bevacizumab and Irinotecan Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 37/60 | 37/57
Other Adverse Events (participants affected / at risk) | 55/60 | 55/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Bevacizumab and Temozolomide) (N=60) | Arm II (Bevacizumab and Irinotecan Hydrochloride) (N=57)
Edema: limb: (Blood and lymphatic system disorders) | 1 | 1
Epistaxis (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 3 | 3
Hemorrhage, GI: Upper GI NOS (Blood and lymphatic system disorders) | 1 | 1
Hemorrhage/bleeding - Other: (Blood and lymphatic system disorders) | 1 | 0
Hemorrhagic stroke (Blood and lymphatic system disorders) | 3 | 1
Intra-abdominal haemorrhage NOS (Blood and lymphatic system disorders) | 1 | 0
Leukopenia NOS (Blood and lymphatic system disorders) | 2 | 6
Lymphopenia (Blood and lymphatic system disorders) | 5 | 5
Neutrophil count (Blood and lymphatic system disorders) | 3 | 4
Platelet count decreased (Blood and lymphatic system disorders) | 7 | 1
Rectal hemorrhage (Blood and lymphatic system disorders) | 1 | 0
Urinary bladder hemorrhage (Blood and lymphatic system disorders) | 1 | 0
Urogenital hemorrhage (Blood and lymphatic system disorders) | 1 | 0
Cardiac General - Other: (Cardiac disorders) | 1 | 0
Hypotension NOS (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Troponin I increased (Cardiac disorders) | 1 | 0
Auditory/ear - Other: (Ear and labyrinth disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 0
Anorexia (Gastrointestinal disorders) | 2 | 0
Colonic perforation (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dehydration (Gastrointestinal disorders) | 0 | 4
Diarrhoea NOS (Gastrointestinal disorders) | 0 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other: (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5
Vomiting NOS (Gastrointestinal disorders) | 0 | 5
Chest pain (General disorders) | 2 | 0
Death NOS (General disorders) | 1 | 1
Disease progression NOS (General disorders) | 5 | 6
Fatigue (General disorders) | 6 | 5
Multi-organ failure (General disorders) | 1 | 0
Pain NOS (General disorders) | 0 | 1
Rhinitis allergic NOS (Immune system disorders) | 0 | 1
Anal infection NOS (Infections and infestations) | 1 | 1
Ano-rectal infection NOS (Infections and infestations) | 0 | 1
Encephalitis NOS (Infections and infestations) | 0 | 1
Febrile neutropenia (Infections and infestations) | 0 | 1
Infection - Other: (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bladder (urinary) (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Colon (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Foreign body (e.g., graft, implant, pro (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Skin (cellulitis) (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Catheter-related (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Colon (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Larynx (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 | 0
Infection with unknown ANC: Upper airway NOS (Infections and infestations) | 0 | 1
Penile infection NOS (Infections and infestations) | 1 | 0
Respiratory tract infection NOS (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Weight decreased (Investigations) | 0 | 2
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 | 1
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 3 | 1
Blood alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 2 | 2
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Metabolic/laboratory - Other: (Metabolism and nutrition disorders) | 3 | 6
Proteinuria (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal/soft tissue - Other: (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Agitation (Nervous system disorders) | 2 | 0
Anxiety (Nervous system disorders) | 1 | 0
Apnoea (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 2
Cerebrospinal fluid leak (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1
Confusional state (Nervous system disorders) | 2 | 1
Convulsions NOS (Nervous system disorders) | 9 | 5
Depression (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 2
Hyperreflexia (Nervous system disorders) | 1 | 4
Memory impairment (Nervous system disorders) | 1 | 0
Mental status changes (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Speech disorder (Nervous system disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary/upper respiratory - Other: (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatology/skin - Other: (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombosis (Vascular disorders) | 3 | 7
Vascular access NOS complication (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Bevacizumab and Temozolomide) (N=60) | Arm II (Bevacizumab and Irinotecan Hydrochloride) (N=57)
Edema: limb: (Blood and lymphatic system disorders) | 16 | 9
Epistaxis (Blood and lymphatic system disorders) | 14 | 10
Hemoglobin (Blood and lymphatic system disorders) | 26 | 23
Hemorrhage/bleeding - Other: (Blood and lymphatic system disorders) | 3 | 0
Hemorrhagic stroke (Blood and lymphatic system disorders) | 3 | 4
Leukopenia NOS (Blood and lymphatic system disorders) | 22 | 21
Lower gastrointestinal hemorrhage (Blood and lymphatic system disorders) | 4 | 2
Lymphopenia (Blood and lymphatic system disorders) | 29 | 30
Neutrophil count (Blood and lymphatic system disorders) | 9 | 18
Platelet count decreased (Blood and lymphatic system disorders) | 30 | 20
Hypertension NOS (Cardiac disorders) | 10 | 12
Hypotension NOS (Cardiac disorders) | 2 | 4
Cushingoid (Endocrine disorders) | 12 | 5
Ocular/visual - Other: (Eye disorders) | 5 | 3
Vision blurred (Eye disorders) | 8 | 3
Abdominal pain NOS (Gastrointestinal disorders) | 6 | 12
Anorexia (Gastrointestinal disorders) | 13 | 9
Constipation (Gastrointestinal disorders) | 13 | 15
Dehydration (Gastrointestinal disorders) | 1 | 5
Diarrhoea NOS (Gastrointestinal disorders) | 11 | 39
Dysgeusia (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 6
Dysphagia (Gastrointestinal disorders) | 3 | 4
Faecal incontinence (Gastrointestinal disorders) | 3 | 0
Gastritis NOS (Gastrointestinal disorders) | 1 | 3
Gastrointestinal - Other: (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 19 | 30
Oral pain (Gastrointestinal disorders) | 2 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 4
Vomiting NOS (Gastrointestinal disorders) | 14 | 17
Fatigue (General disorders) | 39 | 39
Pain - Other: (General disorders) | 2 | 3
Pyrexia (General disorders) | 4 | 4
Rigors (General disorders) | 4 | 2
Syndromes - Other: (General disorders) | 0 | 3
Rhinitis allergic NOS (Immune system disorders) | 1 | 5
Bronchitis NOS (Infections and infestations) | 3 | 1
Respiratory tract infection NOS (Infections and infestations) | 3 | 3
Sinusitis NOS (Infections and infestations) | 1 | 4
Urinary tract infection NOS (Infections and infestations) | 1 | 3
Activated partial thromboplastin time prolonged (Investigations) | 1 | 3
Prothrombin time prolonged (Investigations) | 3 | 1
Weight decreased (Investigations) | 7 | 7
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 21 | 18
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 18 | 12
Blood alkaline phosphatase increased (Metabolism and nutrition disorders) | 9 | 9
Blood amylase increased (Metabolism and nutrition disorders) | 1 | 3
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 5 | 8
Blood bilirubin increased (Metabolism and nutrition disorders) | 6 | 4
Blood creatinine increased (Metabolism and nutrition disorders) | 12 | 7
Gamma-glutamyltransferase increased (Metabolism and nutrition disorders) | 8 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 3
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 34 | 24
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 6
Hypermagnesaemia (Metabolism and nutrition disorders) | 5 | 4
Hypernatremia (Metabolism and nutrition disorders) | 3 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 4 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 21
Hypoglycemia NOS (Metabolism and nutrition disorders) | 8 | 4
Hypokalemia (Metabolism and nutrition disorders) | 10 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 6
Hyponatremia (Metabolism and nutrition disorders) | 10 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 7
Lipase increased (Metabolism and nutrition disorders) | 18 | 3
Metabolic/laboratory - Other: (Metabolism and nutrition disorders) | 10 | 10
Proteinuria (Metabolism and nutrition disorders) | 10 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Gait abnormal NOS (Musculoskeletal and connective tissue disorders) | 5 | 2
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 4 | 12
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 8 | 3
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-upper (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle weakness, generalized or specific area (not due to neuropathy): Right-sided (Musculoskeletal and connective tissue disorders) | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Agitation (Nervous system disorders) | 4 | 3
Anxiety (Nervous system disorders) | 4 | 7
Ataxia (Nervous system disorders) | 7 | 8
Cognitive disorder (Nervous system disorders) | 9 | 5
Confusional state (Nervous system disorders) | 13 | 11
Convulsions NOS (Nervous system disorders) | 13 | 11
Depressed level of consciousness (Nervous system disorders) | 6 | 5
Depression (Nervous system disorders) | 2 | 6
Dizziness (Nervous system disorders) | 8 | 4
Headache (Nervous system disorders) | 19 | 24
Hyperreflexia (Nervous system disorders) | 13 | 7
Memory impairment (Nervous system disorders) | 18 | 11
Mental status changes (Nervous system disorders) | 0 | 4
Neurology - Other: (Nervous system disorders) | 3 | 4
Optic nerve disorder NOS (Nervous system disorders) | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 6 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 7
Personality change (Nervous system disorders) | 4 | 1
Speech disorder (Nervous system disorders) | 16 | 14
Tremor (Nervous system disorders) | 4 | 5
Insomnia (Psychiatric disorders) | 7 | 4
Pollakiuria (Renal and urinary disorders) | 3 | 2
Renal/genitourinary - Other: (Renal and urinary disorders) | 0 | 3
Urinary incontinence (Renal and urinary disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Laryngitis NOS (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pulmonary/upper respiratory - Other: (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Acne NOS (Skin and subcutaneous tissue disorders) | 5 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 3 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2
Sweating increased (Vascular disorders) | 3 | 1
Thrombosis (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less